CLINICAL TRIAL: NCT04973839
Title: Optimizing the Efficacy of Progressive Muscle Relaxation Using Placebo Mechanisms in an Guided and Unguided Online-intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: augment_PMR
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video optimizing expectations before PMR (unguided) (Experimental): watching a video aiming to optimize participants' expectations before undergoing a single PMR session without personal support of the experimenter (unguided)
  Interventions: Behavioral: Video optimizing expectations before PMR (unguided) + Progressive Muscle Relaxation (PMR)
- Video optimizing expectations before PMR (guided) (Experimental): watching a video aiming to optimize participants' expectations before undergoing a single PMR session with the personal support of the experimenter (guided)
  Interventions: Behavioral: Video optimizing expectations before PMR (guided) + Progressive Muscle Relaxation (PMR)
- Neutral video before PMR (unguided) (Active Comparator): watching a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session without personal support of the experimenter (unguided),
  Interventions: Behavioral: Neutral video before PMR (unguided) + Progressive Muscle Relaxation (PMR)
- Neutral video before PMR (guided) (Active Comparator): watching a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session with the personal support of the experimenter (guided)
  Interventions: Behavioral: Neutral video before PMR (guided)+ Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Behavioral: Video optimizing expectations before PMR (unguided) + Progressive Muscle Relaxation (PMR) — Participants watch a video aiming to optimize participants' expectations before undergoing a single PMR session without personal support of the experimenter (unguided). The PMR session involves learning to monitor tension in each specific muscle group in the body by deliberately inducing tension in each group. This tension is then released, with attention paid to the contrast between tension and relaxation.
  Arms: Video optimizing expectations before PMR (unguided)
Behavioral: Video optimizing expectations before PMR (guided) + Progressive Muscle Relaxation (PMR) — Participants watch a video aiming to optimize participants' expectations before undergoing a single PMR session with the personal support of the experimenter (guided). The PMR session involves learning to monitor tension in each specific muscle group in the body by deliberately inducing tension in each group. This tension is then released, with attention paid to the contrast between tension and relaxation.
  Arms: Video optimizing expectations before PMR (guided)
Behavioral: Neutral video before PMR (unguided) + Progressive Muscle Relaxation (PMR) — Participants watch a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session without personal support of the experimenter (unguided). The PMR session involves learning to monitor tension in each specific muscle group in the body by deliberately inducing tension in each group. This tension is then released, with attention paid to the contrast between tension and relaxation.
  Arms: Neutral video before PMR (unguided)
Behavioral: Neutral video before PMR (guided)+ Progressive Muscle Relaxation (PMR) — Participants watch a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session with the personal support of the experimenter (guided).The PMR session involves learning to monitor tension in each specific muscle group in the body by deliberately inducing tension in each group. This tension is then released, with attention paid to the contrast between tension and relaxation.
  Arms: Neutral video before PMR (guided)

SUMMARY:
This study aims to determine whether a brief video aiming to optimize expectations regarding the effectiveness of progressive muscle relaxation (PMR) can enhance the efficacy of a PMR compared to a neutral video control group in an online intervention. Another aim is to assess whether this effect will be moderated by the degree of human support (guided or unguided intervention).

DETAILED DESCRIPTION:
This study aims to determine whether a brief video aiming to optimize expectations regarding the effectiveness of progressive muscle relaxation (PMR) can enhance the efficacy of a PMR session compared to a neutral video control group in an online intervention. Another aim is to assess whether this effect will be moderated by the degree of human support (guided or unguided intervention). After the baseline assessment, participants are randomized to one of 4 possible intervention groups: i) watching a video aiming to optimize participants' expectations before undergoing a single PMR session without personal support of the experimenter (unguided), ii) watching a video aiming to optimize participants' expectations before undergoing a single PMR session with the personal support of the experimenter (guided), iii) watching a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session without personal support of the experimenter (unguided), or iv) watching a neutral video (not aiming to optimize participants' expectations) before undergoing a single PMR session with the personal support of the experimenter (guided). In a pre-posttest design, the subjective stress levels of the participants in the for groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* fluency in the German language to provide informed consent

Exclusion Criteria:

* muscle disease, muscle cramps, acute psychosis, acute trauma responses, or another chronic somatic illness
* Mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate how stressed they feel at the moment at two time points (baseline and after the PMR intervention) on a questionnaire (VAS: item ranges from 0 (not stressed at all) - 100 (very stressed). Change scores are calculated (post- minus pre-scores). More negative change scores are better since it indicates a stronger stress reduction (maximum reduction: -100). Higher positive change scores are worse since this indicates an increase in perceived stress (maximum increase: +100). Range of change scores: -100 - +100).

SECONDARY OUTCOMES:
Change in positive affect | Change from pre (baseline) to post scores (30 minutes later)
  Participants are asked to rate adjectives regarding their current mood (positive and negative) at two time points (baseline and after the PMR intervention) on a questionnaire. Change scores are calculated (post- minus pre-scores). Instrument: Positive and Negative Affect Scale (PANAS) by Watson, Clark, and Tellegen (1988) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Range for sum score of positive/negative affect: 10-50. For positive affect higher scores are better; for negative affect lower scores are better.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided